CLINICAL TRIAL: NCT06910865
Title: Study of the Radio-clinical Correlation of Endolymphatic Hydrops
Acronym: CRHE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9306
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Endolymphatic Hydrops
Keywords: Endolymphatic Hydrops
MeSH Terms: conditions — Endolymphatic Hydrops

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In patients presenting with symptoms of endolymphatic hydrops, signs of vestibular dilation are often found on MRI. Some patients present with these radiological signs without vestibular clinical signs, or signs other than those of hydrops. No study has yet investigated the radiological-clinical correlation of endolymphatic hydrops by selecting patients based on their imaging findings and then comparing them to the symptoms presented.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (≥18 years)
* Subject presenting vestibular dilation on MRI

Exclusion Criteria:

* Subjects who have expressed opposition to the reuse of their data for scientific research purposes.
* Subjects under legal protection
* Subjects under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subject (≥18 years) presenting vestibular dilation on MRI
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Nystagmus observed on videonystagmoscopy | Up to 1 year
  Nystagmus observed on videonystagmoscopy:
  * Unidirectional or multidirectional
  * Direction
  * Exhaustible or not
  * Perceptible or not

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et de Chirurgie Cervico-faciale - CHU de Strasbourg - France, Strasbourg, France